CLINICAL TRIAL: NCT04741308
Title: The Effect of Cognitive Behavior Therapy (CBT) on Psychological Status and Immune Function of Colorectal Cancer Patients Undergoing Chemotherapy.
Brief Title: Cognitive Behavior Therapy (CBT) and Psychological Status and Immune Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Yuan Shen, MD, PhD, Chief of Psychiatry, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: dsyy006
Record Dates: First submitted 2021-01-27; First posted 2021-02-05 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer; Cognitive Behavior Therapy; Immune Function
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT group (Experimental): Patients randomly assigned to CBT group will receive 8 times of CBT treatment during chemotherapy.
  Interventions: Behavioral: cognitive behavior therapy
- non-CBT group (No Intervention): Patients randomly assigned to non-CBT group will receive four sessions of health education in a month after surgery.
  Each session will last 1 hour, including lectures and Q&A . The content of each session is different, including: diagnosis and treatment of colorectal cancer, adverse reactions and management of chemotherapy, nutritional support during chemotherapy and physical exercise during chemotherapy.

INTERVENTIONS:
Behavioral: cognitive behavior therapy — The CBT intervention is a 8-times group-based intervention that meets 2-3 weeks.Each session will be performed during chemotherapy and will last for 60 min, including 45 min cognitive behavior therapy and 15 min relaxation training.Our CBT intervention is designed to be conducted in groups of 3 to 6 patients led by two group facilitators. Group leaders will: guide participants relaxation training, develop a supportive group environment, encourage emotional expression, assist participants develop a sense of self-confidence, identify maladaptive coping and encourage adaptive coping responses.
  Arms: CBT group

SUMMARY:
To explore the effect of CBT on psychological status of colorectal cancer patients undergoing chemotherapy. To explore the effect of CBT on immune function of colorectal cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Cancer patients undergoing chemotherapy are often subjected to considerable psychological stress. CBT is considered as one of the effective methods to relieve stress. CBT is effective in alleviating depression and anxiety, but the effect of CBT on cognitive and immune function in patients with colorectal cancer undergoing chemotherapy remains uninvestigated.

ELIGIBILITY:
Inclusion Criteria:

1.18≤age≤75; 2.Being scheduled to undergo colorectal cancer surgery; 3.Being able to complete all the assessment.

Exclusion Criteria:

1. Having a history of tumor, mental disorders(including dementia), brain trauma or other cerebral diseases;
2. Having severe depression and anxiety currently;
3. Having alcohol dependence or other substance dependence;
4. Having serious physical illness;
5. Participating in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline stress perception at follow-up. | Baseline and follow-up ( immediately after intervention, 3 months and 6 months after intervention).
  Stress perception will be assessed by Perceived Stress Scale (PSS-10). The sum score of PSS-10 ranges from 0 to 40. Higher scores mean a worse outcome.
Change from baseline depressionat at follow-up. | Baseline and follow-up ( immediately after intervention, 3 months and 6 months after intervention).
  Depression will be assessed by Patient Health Questionnaire (PHQ-9). The sum score of PHQ-9 ranges from 0 to 27. Higher scores mean a worse outcome.
Change from baseline anxiety at follow-up. | Baseline and follow-up ( immediately after intervention, 3 months and 6 months after intervention).
  Anxiety will be assessed by Generalized Anxiety Disorder (GAD-7). The sum score of GAD-7 ranges from 0 to 21. Higher scores mean a worse outcome.
Change from baseline cognitive function at follow-up. | Baseline and follow-up ( immediately after intervention, 3 months and 6 months after intervention).
  Cognitive function will be assessed by Mini-mental State Examination (MMSE), Hopkins Verbal Learning Test-Revised, Digit Span Test, Digit-symbol Test and Trail Making Test.
Change from baseline immune function at follow-up. | Baseline and follow-up ( immediately after intervention, 3 months and 6 months after intervention).
  Immune function assessment includes cytokine levels (IL-1α, IL-1β, IL-6, IL-8, TNF-α, TNF-β, CRP) and immune cell levels (CD4+T cell, CD8+T cell, natural killer, monocytes, B cell).

SECONDARY OUTCOMES:
Change from baseline quality of life of patient at follow-up. | Baseline and follow-up ( immediately after intervention, 3 months and 6 months after intervention).
  It will be assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer 29 (EORTC QLQ-CR29).
Change from baseline sleep quality at follow-up. | Baseline and follow-up ( immediately after intervention, 3 months and 6 months after intervention).
  It will be assessed by Pittsburgh sleep quality index (PSQI).
Change from baseline self efficacy at follow-up. | Baseline and follow-up ( immediately after intervention, 3 months and 6 months after intervention).
  It will be assessed by General Self Efficacy (GSES). The sum score of General Self Efficacy ranges from 10 to 40. Higher scores mean a better outcome.
Social support | Baseline.
  It will be assessed by Social Support Rating Scale (SSRS). The sum score of Social Support Rating Scale ranges from 12 to 66. Higher scores mean a better outcome.
Change from baseline chemotherapy response at follow-up. | Baseline and follow-up ( immediately after intervention, 3 months and 6 months after intervention).
  It will be evaluated by M.D. Anderson Symptom Inventory-Gastrointestinal Cancer Module (MDASI-GI).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang M, Xu Y, Shi J, Zhuang C, Zhuang Y, Li J, Cashin PH. The effect of cognitive behavioral therapy on chemotherapy-induced side effects and immune function in colorectal cancer patients undergoing chemotherapy: study protocol for a randomized controlled trial. J Gastrointest Oncol. 2023 Aug 31;14(4):1869-1877. doi: 10.21037/jgo-23-625. Epub 2023 Aug 30. PMID 37720456